CLINICAL TRIAL: NCT03041311
Title: Phase 2 Study of Carboplatin, Etoposide, and Atezolizumab With or Without Trilaciclib in Patients With Untreated Extensive-Stage Small Cell Lung Cancer (SCLC)
Brief Title: Carboplatin, Etoposide, and Atezolizumab With or Without Trilaciclib (G1T28), a CDK4/6 Inhibitor, in Extensive-Stage SCLC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: G1 Therapeutics, Inc. (Industry)
Collaborators: Roche-Genentech (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: G1T28-05; 2017-000358-20 (EudraCT Number)
Record Dates: First submitted 2017-02-01; First posted 2017-02-02 (Estimated); Results first posted 2022-05-06 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Small Cell Lung Cancer
Keywords: Small Cell Lung Cancer; CDK4/6 Inhibitor; Immune Checkpoint Inhibitor
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — trilaciclib; Carboplatin; Etoposide; atezolizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- trilaciclib+etoposide/carboplatin/atezolizumab (Experimental): Induction: Patients received trilaciclib 240 mg/m² administered intravenously (IV) once daily prior to E/P/A on Days 1, 2 and 3 of each 21-day E/P/A therapy cycle (up to 4 cycles in total). Etoposide 100 mg/m² was administered IV daily on Days 1, 2, and 3 of each 21-day cycle. Carboplatin was administered on Day 1 of each 21-day cycle using the Calvert formula with a target area under the concentration-time curve (AUC) = 5 milligrams per milliliter per minute (mg/mL/min) to calculate the dose. Atezolizumab 1200 mg was administered as an IV infusion on Day 1 of each 21-day cycle.
  Maintenance: Following the induction phase, patients received maintenance atezolizumab at a dose of 1200 mg on Day 1 of every 21-day cycle until disease progression, unacceptable toxicity or discontinuation by the patient or investigator.
  Interventions: Drug: Trilaciclib; Drug: Carboplatin; Drug: Etoposide; Drug: Atezolizumab
- placebo+etoposide/carboplatin/atezolizumab (Experimental): Induction: Patients received placebo administered IV once daily prior to E/P/A on Days 1, 2 and 3 of each 21-day E/P/A therapy cycle (up to 4 cycles in total). Etoposide 100 mg/m² was administered IV daily on Days 1, 2, and 3 of each 21-day cycle. Carboplatin was be administered on Day 1 of each 21-day cycle using the Calvert formula with a target AUC = 5 mg/mL/min to calculate the dose. Atezolizumab 1200 mg was administered as an IV infusion on Day 1 of each 21-day cycle.
  Maintenance: Following the induction phase, patients received maintenance atezolizumab at a dose of 1200 mg on Day 1 of every 21-day cycle until disease progression, unacceptable toxicity or discontinuation by the patient or investigator.
  Interventions: Drug: Placebo; Drug: Carboplatin; Drug: Etoposide; Drug: Atezolizumab

INTERVENTIONS:
Drug: Trilaciclib — Trilaciclib IV
  Other Names: G1T28
  Arms: trilaciclib+etoposide/carboplatin/atezolizumab
Drug: Placebo — Placebo IV
  Arms: placebo+etoposide/carboplatin/atezolizumab
Drug: Carboplatin — Carboplatin IV
  Other Names: Paraplatin
Drug: Etoposide — Etoposide IV
  Other Names: VP-16
Drug: Atezolizumab — Atezolizumab IV
  Other Names: Tecentriq

SUMMARY:
This was a study to investigate the potential clinical benefit of trilaciclib (G1T28) in preserving the bone marrow and the immune system, and enhancing antitumor efficacy when administered with carboplatin, etoposide, and atezolizumab (E/P/A) therapy in first line treatment for patients with newly diagnosed extensive-stage SCLC.

The study was a randomized, double-blinded, placebo-controlled design. Approximately, 100 patients were randomized to trilaciclib + E/P/A or placebo + E/P/A in the study.

DETAILED DESCRIPTION:
The posted results represent the final results from Study G1T28-05, a Phase 2 study of carboplatin, etoposide, and atezolizumab with or without trilaciclib (G1T28) in patients with untreated extensive-stage small cell lung cancer (SCLC).

The final myelopreservation efficacy results are from database lock 1 (data cut-off [DCO] 17 Aug 2018). The final anti-tumor efficacy data (BOR, DOR, PFS) are from a second database lock 2 (DCO 28 June 2019) that occurred to support the trilaciclib New Drug Application (NDA). Final overall survival and safety data are reported from the final study database lock (DCO 11 Dec 2020, last patient last visit date of 29 October 2020).

Please note the last patient last visit date description above which is recorded as the study completion date. Following the last patient last visit, the final database lock occurred a few weeks later which accounts for the discrepancy between the study completion date and the reported assessment time frames.

ELIGIBILITY:
Key Inclusion Criteria:

* Male or female subjects aged ≥18 years
* Unequivocally confirmed diagnosis of SCLC by histology or cytology, preferably including the presence of neuroendocrine features by immunohistochemistry
* Extensive-stage SCLC
* At least 1 target lesion that is measurable by Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1
* Adequate organ function
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 - 2
* Predicted life expectancy of ≥3 months
* Able to understand and sign an informed consent

Exclusion Criteria:

* Limited-stage SCLC
* Prior chemotherapy for limited or extensive-stage SCLC
* Prior treatment with immunotherapies including but not limited to cluster of differentiation 137 agonists or immune checkpoint blockade therapies (such as anti-programmed cell death protein 1 (PD-1), anti-programmed death-ligand 1(PD-L1), and cytotoxic T-lymphocyte-associated protein 4 (CTLA-4) therapeutic antibodies).
* Presence of symptomatic brain metastases requiring immediate treatment with radiation therapy or steroids.
* Malignancies other than SCLC within 3 years prior to randomization, with the exception of those with negligible risk of metastasis or death treated with expected curative outcome
* History of idiopathic pulmonary fibrosis, organizing pneumonia, drug induced pneumonitis, idiopathic pneumonitis, or evidence of active pneumonitis on screening chest CT scan
* Active, known, suspected autoimmune disease requiring systemic treatment in the past 2 years
* Uncontrolled ischemic heart disease or uncontrolled symptomatic congestive heart failure
* Known history of stroke or cerebrovascular accident within 6 months prior to enrollment
* Serious active infection at the time of enrollment
* Psychiatric illness/social situations that would limit study compliance
* Other uncontrolled serious chronic disease or conditions that in the investigator's opinion could affect compliance or follow-up in the protocol
* Known human immunodeficiency virus, known active hepatitis B, or hepatitis C
* Radiotherapy to any site or radiotherapy within 2 weeks prior to enrollment
* Receipt of any investigational medication within 4 weeks prior to enrollment
* Administration of attenuated vaccine within 4 weeks before enrollment or anticipation that such a live attenuated vaccine will be required during the study
* Influenza vaccination should be given during influenza season only (approx. Oct to March). Patients must not receive live, attenuated influenza vaccine (eg, FluMist) within 4 weeks prior to enrollment at any time during the study, and at least 5 months after the last dose of atezolizumab.
* Patients with a condition requiring systemic treatment with either corticosteroids ( > 10 mg daily prednisone equivalents) or other immunosuppressive medications (including but not limited to cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor agents) within 14 days of study drug administration. Inhaled or topical steroids ad adrenal replacement dosed > 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease.
* Hypersensitivity to any of the components of the formulation of etoposide or etoposide phosphate
* Hypersensitivity to carboplatin or other platinum-containing compounds or to mannitol
* History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins
* Known hypersensitivity to Chinese hamster ovary cell products or other recombinant human antibodies
* Legal incapacity or limited legal capacity
* Pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2017-06-29 (Actual); Primary Completion 2018-08-17 (Actual); Study Completion 2020-10-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Contact, Study Director — G1 Therapeutics, Inc.
Locations (45):
- United States (23):
  - Beverly Hills Cancer Center, Beverly Hills, California
  - St. Jude Heritage Healthcare, Fullerton, California
  - Loma Linda University, Loma Linda, California
  - UCLA Medical Center - Santa Monica Hematology And Oncology, Santa Monica, California
  - Redwood Regional Medical Group (RRMG) - Fountain Grove, Santa Rosa, California
  - Singing River Health System, Whittier, California
  - Piedmont Cancer Institute, Atlanta, Georgia
  - Northside Hospital - Georgia Cancer Specialists, Atlanta, Georgia
  - Joliet Oncology-Hematology Associates, Joliet, Illinois
  - Horizon Oncology Center, Lafayette, Indiana
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - St. Louis Cancer Care, LLP, North County, Bridgeton, Missouri
  - The Alvin J. Siteman Cancer Center - Center for Advanced Med, St Louis, Missouri
  - Summit Medical Group, P.A., Morristown, New Jersey
  - Northern Westchester Hospital, Mount Kisco, New York
  - Trinity Health - Trinity CancerCare Center, Minot, North Dakota
  - Oklahoma University - Peggy and Charles Stephenson Cancer Center, Oklahoma City, Oklahoma
  - Gibbs Cancer Center, Spartanburg, South Carolina
  - Valley Cancer Associates, Harlingen, Texas
  - Millennium Oncology, Houston, Texas
  - Virginia Cancer Specialists, Arlington, Virginia
  - Blue Ridge Cancer Care, Blacksburg, Virginia
  - Fort Belvoir Community Hospital, Fort Belvoir, Virginia
- Bulgaria (3):
  - Complex Oncology Center - Burgas, Burgas
  - Multiprofile Hospital for Active Treatment "Serdika", Sofia, Sofia
  - Multiprofile Hospital for Active Treatment "Serdika", Sofia
- East Tallinn Central Hospital Ltd., Clinic of Internal Medicine, Center for Oncology, Tallinn, Estonia
- France (2):
  - CHU Caen De La Côte De Nacre, Caen
  - Centre Oscar Lambret, Lille
- Latvia (2):
  - Daugavpils Regional Hospital, Department of Oncology, Daugavpils
  - Pauls Stradiņš Clinical University Hospital, Oncology Clinic, Riga
- Spain (11):
  - Hospital Universitario Son Espases, Palma, Balearic Islands
  - Hospital Teresa Herrera, A Coruña, La Coruña
  - Hospital Universitario Puerta de Hierro Majadahonda, Majadahonda, Madrid
  - Hospital Clínico, San Carlos, Madrid
  - H.U. Quirón Dexeus, Hospital Universitario, Barcelona
  - Hospital Clinic de Barcelona- Servicio de Oncología Médica, Barcelona
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital 12 de Octubre, Madrid
  - H. Donostia, Hospital Donostia- Servicio de Oncología, San Sebastián
  - Hospital Universitario Ntra. Sra. de Valme, Seville
  - Hospital Arnau de Vilanova, Valencia
- Ukraine (3):
  - Chernivtsi Regional Clinical Oncology Center, Chernivtsi
  - Dnipropetrovsk City Multispecialty Clinical Hospital #4, Dnipro
  - Lviv State Regional Treatment and Diagnostics Oncology Center, Lviv

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Daniel D, Kuchava V, Bondarenko I, Ivashchuk O, Reddy S, Jaal J, Kudaba I, Hart L, Matitashvili A, Pritchett Y, Morris SR, Sorrentino JA, Antal JM, Goldschmidt J. Trilaciclib prior to chemotherapy and atezolizumab in patients with newly diagnosed extensive-stage small cell lung cancer: A multicentre, randomised, double-blind, placebo-controlled Phase II trial. Int J Cancer. 2021 May 15;148(10):2557-2570. doi: 10.1002/ijc.33453. Epub 2021 Jan 12. PMID 33348420
- [Background] Weiss J, Goldschmidt J, Andric Z, Dragnev KH, Gwaltney C, Skaltsa K, Pritchett Y, Antal JM, Morris SR, Daniel D. Effects of Trilaciclib on Chemotherapy-Induced Myelosuppression and Patient-Reported Outcomes in Patients with Extensive-Stage Small Cell Lung Cancer: Pooled Results from Three Phase II Randomized, Double-Blind, Placebo-Controlled Studies. Clin Lung Cancer. 2021 Sep;22(5):449-460. doi: 10.1016/j.cllc.2021.03.010. Epub 2021 Mar 26. PMID 33895103
- [Derived] Abraham I, Onyekwere U, Deniz B, Moran D, Chioda M, MacDonald K, Huang H. Trilaciclib and the economic value of multilineage myeloprotection from chemotherapy-induced myelosuppression among patients with extensive-stage small cell lung cancer treated with first-line chemotherapy. J Med Econ. 2021 Nov;24(sup1):71-83. doi: 10.1080/13696998.2021.2014163. PMID 34873975
- [Derived] Zeng R, Liu F, Fang C, Yang J, Luo L, Yue P, Gao B, Dong Y, Xiang Y. PIV and PILE Score at Baseline Predict Clinical Outcome of Anti-PD-1/PD-L1 Inhibitor Combined With Chemotherapy in Extensive-Stage Small Cell Lung Cancer Patients. Front Immunol. 2021 Oct 29;12:724443. doi: 10.3389/fimmu.2021.724443. eCollection 2021. PMID 34777341
- [Derived] Hussein M, Maglakelidze M, Richards DA, Sabatini M, Gersten TA, Lerro K, Sinielnikov I, Spira A, Pritchett Y, Antal JM, Malik R, Beck JT. Myeloprotective Effects of Trilaciclib Among Patients with Small Cell Lung Cancer at Increased Risk of Chemotherapy-Induced Myelosuppression: Pooled Results from Three Phase 2, Randomized, Double-Blind, Placebo-Controlled Studies. Cancer Manag Res. 2021 Aug 9;13:6207-6218. doi: 10.2147/CMAR.S313045. eCollection 2021. PMID 34408488
- [Derived] Ferrarotto R, Anderson I, Medgyasszay B, Garcia-Campelo MR, Edenfield W, Feinstein TM, Johnson JM, Kalmadi S, Lammers PE, Sanchez-Hernandez A, Pritchett Y, Morris SR, Malik RK, Csoszi T. Trilaciclib prior to chemotherapy reduces the usage of supportive care interventions for chemotherapy-induced myelosuppression in patients with small cell lung cancer: Pooled analysis of three randomized phase 2 trials. Cancer Med. 2021 Sep;10(17):5748-5756. doi: 10.1002/cam4.4089. Epub 2021 Aug 18. PMID 34405547

RESULTS

PARTICIPANT FLOW:
Groups:
- Trilaciclib+Etoposide/Carboplatin/Atezolizumab: Induction: Patients received trilaciclib 240 mg/m² administered IV once daily prior to E/P/A on Days 1, 2 and 3 of each 21-day E/P/A therapy cycle (up to 4 cycles in total). Etoposide 100 mg/m² was administered IV daily on Days 1, 2, and 3 of each 21-day cycle. Carboplatin was administered on Day 1 of each 21-day cycle using the Calvert formula with a target AUC = 5 mg/mL/min to calculate the dose. Atezolizumab 1200 mg was administered as an IV infusion on Day 1 of each 21-day cycle.
  Maintenance: Following the induction phase, patients received maintenance atezolizumab at a dose of 1200 mg on Day 1 of every 21-day cycle until disease progression, unacceptable toxicity, or discontinuation by the patient or investigator.
- Placebo+Etoposide/Carboplatin/Atezolizumab: Induction: Patients received placebo administered IV once daily prior to E/P/A on Days 1, 2 and 3 of each 21-day E/P/A therapy cycle (up to 4 cycles in total). Etoposide 100 mg/m² was administered IV daily on Days 1, 2, and 3 of each 21-day cycle. Carboplatin was administered on Day 1 of each 21-day cycle using the Calvert formula with a target AUC = 5 mg/mL/min to calculate the dose. Atezolizumab 1200 mg was administered as an IV infusion on Day 1 of each 21-day cycle.
  Maintenance: Following the induction phase, patients received maintenance atezolizumab at a dose of 1200 mg on Day 1 of every 21-day cycle until disease progression, unacceptable toxicity, or discontinuation by the patient or investigator.
Period: Overall Study
Arm/Group | Trilaciclib+Etoposide/Carboplatin/Atezolizumab | Placebo+Etoposide/Carboplatin/Atezolizumab
Started | 54 | 53
Completed | 0 | 0
Not Completed | 54 | 53
Not completed — Death | 39 | 42
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 8 | 5
Not completed — Sponsor Terminated Study | 2 | 4
Not completed — Disease Progression | 3 | 1
Not completed — Randomized in error, did not receive drug | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Trilaciclib+Etoposide/Carboplatin/Atezolizumab: Induction: Patients received trilaciclib 240 mg/m² administered IV once daily on Days prior to E/P/A 1, 2 and 3 of each 21-day E/P/A therapy cycle (up to 4 cycles in total). Etoposide 100 mg/m² was administered IV daily on Days 1, 2, and 3 of each 21-day cycle. Carboplatin was administered on Day 1 of each 21-day cycle using the Calvert formula with a target AUC = 5 mg/mL/min to calculate the dose. Atezolizumab 1200 mg was administered as an IV infusion on Day 1 of each 21-day cycle.
  Maintenance: Following the induction phase, patients received maintenance atezolizumab at a dose of 1200 mg on Day 1 of every 21-day cycle until disease progression, unacceptable toxicity, or discontinuation by the patient or investigator.
- Placebo+Etoposide/Carboplatin/Atezolizumab: Induction: Patients received placebo administered IV once daily prior to E/P/A on Days 1, 2 and 3 of each 21-day E/P/A therapy cycle (up to 4 cycles in total). Etoposide 100 mg/m² was administered IV daily on Days 1, 2, and 3 of each 21-day cycle. Carboplatin was administered on Day 1 of each 21-day cycle using the Calvert formula with a target AUC = 5 mg/mL/min to calculate the dose. Atezolizumab 1200 mg was administered as an IV infusion on Day 1 of each 21-day cycle.
  Maintenance: Following the induction phase, patients received maintenance atezolizumab at a dose of 1200 mg on Day 1 of every 21-day cycle until disease progression, unacceptable toxicity or discontinuation by the patient or investigator.
- Total: Total of all reporting groups
Arm/Group | Trilaciclib+Etoposide/Carboplatin/Atezolizumab | Placebo+Etoposide/Carboplatin/Atezolizumab | Total
Number analyzed (Participants) | 54 | 53 | 107
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 27 | 27 | 54
  >=65 years | 27 | 26 | 53
Age, Continuous [Mean (Standard Deviation); unit: years] | 63 (8.4) | 64 (8.3) | 64 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 19 | 32
  Male | 41 | 34 | 75
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 53 | 51 | 104
  Black or African American | 0 | 1 | 1
  Native Hawaiian or Pacific Islander | 1 | 0 | 1
  Other | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  Latvia | 3 | 3 | 6
  United States | 20 | 22 | 42
  Ukraine | 11 | 8 | 19
  Bulgaria | 6 | 7 | 13
  France | 0 | 2 | 2
  Estonia | 2 | 3 | 5
  Spain | 1 | 3 | 4
  Georgia | 11 | 5 | 16
Body Weight at Screening [Mean (Standard Deviation); unit: kg] | 79.2 (17.32) | 72.4 (14.42) | 75.8 (16.25)
Height at Screening [Mean (Standard Deviation); unit: cm] | 171.1 (7.62) | 168.6 (10.21) | 169.9 (9.04)
BMI at Screening [Mean (Standard Deviation); unit: kg/m²] | 27.10 (5.907) | 25.45 (4.618) | 26.28 (5.347)
Body Surface Area (m²) at Screening [Mean (Standard Deviation); unit: m²] | 1.91 (0.198) | 1.82 (0.205) | 1.86 (0.205)
ECOG Performance Status [Count of Participants; unit: Participants] — The publicly available Easter Cooperative Oncology Group (ECOG) Performance Status Scale was utilized to assess patient level of functioning. Increasing numbers indicate worse outcomes.
  GRADE ECOG PERFORMANCE STATUS 0 Fully active, able to carry on all pre-disease performance without restriction
  1. Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work
  2. Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours
  Participants
    0-1 | 46 | 46 | 92
    2 | 8 | 7 | 15

OUTCOME MEASURES:

1. Primary Outcome: Duration of Severe (Grade 4) Neutropenia in Cycle 1
Description: Duration of severe neutropenia (DSN; days) was defined as the number of days from the date of the first absolute neutrophil count (ANC) value of <0.5 × 10⁹/L observed between start of cycle and end of cycle to the date of the first ANC value ≥0.5 × 10⁹/L that met the following criteria: (1) occurred after the ANC value of <0.5 × 10⁹/L and (2) no other ANC values <0.5 × 10⁹/L occurred between this day and end of cycle. DSN was set to 0 for patients who did not experience severe neutropenia in a cycle, including those that were randomized and not treated. Data from unscheduled visits and the actual assessment date (rather than visit date) were included in the derivation.
Time Frame: Evaluated for Cycle 1 of the Induction Period (i.e., from randomization to the end of Cycle 1, each cycle = 21 days).
Population: Intent-to-treat (ITT) analysis set included all randomized patients. Analysis using the ITT analysis set were conducted on the basis of the randomly assigned treatment.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Trilaciclib+Etoposide/Carboplatin/Atezolizumab | Placebo+Etoposide/Carboplatin/Atezolizumab
Number analyzed (Participants) | 54 | 53
days | 0 (1.0) | 4 (4.7)
Statistical Analysis 1: Comparison: Trilaciclib+Etoposide/Carboplatin/Atezolizumab vs Placebo+Etoposide/Carboplatin/Atezolizumab; Treatment difference was evaluated using a nonparametric analysis of covariance (ANCOVA). The nonparametric ANCOVA included study baseline ANC value as covariate, stratification factors of ECOG performance status (0 to 1 versus 2) and brain metastases (Yes versus No), and treatment as a fixed effect; Test type: Superiority; p < 0.0001, non-parametric ANCOVA — A Hochberg-based gatekeeping procedure was used to control the global familywise error rate across the multiple null hypotheses (for 2 primary and 3 key secondary endpoints) in a strong sense at a 1-sided 0.025 level; Hochberg-based gatekeeping procedure

2. Primary Outcome: Number of Participants With at Least 1 Occurrence of Severe (Grade 4) Neutropenia
Description: The occurrence of severe (Grade 4) neutropenia (SN) was a binary variable. If a patient had at least 1 absolute neutrophil count value <0.5 × 10^9/L during the Induction Period, the patient was assigned as Yes to the occurrence of SN; otherwise, it was No.
Time Frame: Induction Period. From date of randomization, 21 day treatment cycles up to a maximum of 4 cycles or until (if earlier) disease progression, unacceptable toxicity, or discontinuation by the patient or investigator, assessed up to a maximum of 409 days.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Placebo+Etoposide/Carboplatin/Atezolizumab: Induction: Patients received placebo administered IV once daily prior to E/P/A on Days 1, 2 and 3 of each 21-day E/P/A therapy cycle (up to 4 cycles in total). Etoposide 100 mg/m² was be administered IV daily on Days 1, 2, and 3 of each 21-day cycle. Carboplatin was administered on Day 1 of each 21-day cycle using the Calvert formula with a target AUC = 5 mg/mL/min to calculate the dose. Atezolizumab 1200 mg was administered as an IV infusion on Day 1 of each 21-day cycle.
  Maintenance: Following the induction phase, patients received maintenance atezolizumab at a dose of 1200 mg on Day 1 of every 21-day cycle until disease progression, unacceptable toxicity, or discontinuation by the patient or investigator.
Arm/Group | Trilaciclib+Etoposide/Carboplatin/Atezolizumab | Placebo+Etoposide/Carboplatin/Atezolizumab
Number analyzed (Participants) | 54 | 53
Participants | 1 | 26
Statistical Analysis 1: Comparison: Trilaciclib+Etoposide/Carboplatin/Atezolizumab vs Placebo+Etoposide/Carboplatin/Atezolizumab; The occurrence of SN was a binary variable. Treatment group difference was analyzed using a modified Poisson regression model to account for the variable duration of the Induction Period for each patient. The model included baseline ANC count as a covariate, the stratification factors of ECOG performance status (0 to1 vs. 2) and brain metastases (Yes vs. No), and treatment as a fixed effect. The logarithm transformation of # of Induction cycles was included as an offset variable in the modeling; Test type: Superiority; p < 0.0001, Modified Poisson — [p-value comment as in outcome 1, analysis 1]; Hochberg-based gatekeeping procedure

3. Secondary Outcome: All-Cause Dose Reductions
Description: Dose reductions are not permitted for trilaciclib or atezolizumab. Dose reductions for E/P are derived from changes in the protocol-specified dose on the dosing page and correspond to the reductions for toxicity specified in the protocol. No more than 2 dose reductions of E/P in total were allowed for any patient. Simultaneous reduction in the doses of etoposide and carboplatin were counted as 1 dose reduction.
Time Frame: Induction Period. From date of randomization, 21 day treatment cycles to a maximum of 4 cycles or until (if earlier) disease progression, unacceptable toxicity, or discontinuation by the patient or investigator, assessed up to a maximum of 409 days.
Population: as for outcome 1
Measure: Number; unit: Events/Cycle
Arm/Group | Trilaciclib+Etoposide/Carboplatin/Atezolizumab | Placebo+Etoposide/Carboplatin/Atezolizumab
Number analyzed (Participants) | 54 | 53
Events/Cycle | 0.021 | 0.085
Statistical Analysis 1: Comparison: Trilaciclib+Etoposide/Carboplatin/Atezolizumab vs Placebo+Etoposide/Carboplatin/Atezolizumab; Test type: Superiority; p = 0.0195, negative binomial regression — [p-value comment as in outcome 1, analysis 1]; Hochberg-based gatekeeping procedure

4. Secondary Outcome: Number of Participants With at Least 1 Occurrence of RBC Transfusion on/After Week 5 (Proportion of Patients)
Description: For this endpoint, the occurrence during the Induction Period was defined as a binary variable (Yes or No); Yes, if total number of events ≥1 was observed, No for other scenarios. If a patient did not have an event, a value of 0 was assigned to that patient. Each red blood cell transfusion with a unique start date on/after Week 5 on study during the Induction was defined as a separate event.
Time Frame: Induction Period. From date of randomization, 21 day treatment cycles to a maximum of 4 cycles or until (if earlier) disease progression, unacceptable toxicity, or discontinuation by the patient or investigator, assessed up to a maximum of 374 days.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Trilaciclib+Etoposide/Carboplatin/Atezolizumab | Placebo+Etoposide/Carboplatin/Atezolizumab
Number analyzed (Participants) | 54 | 53
Participants | 7 | 11
Statistical Analysis 1: Comparison: Trilaciclib+Etoposide/Carboplatin/Atezolizumab vs Placebo+Etoposide/Carboplatin/Atezolizumab; Treatment group difference was analyzed using a modified Poisson regression model. The model included baseline hemoglobin as a covariate, the stratification factors of ECOG performance status (0 to 1 versus 2) and brain metastases (Yes versus No) and treatment as a fixed effect. The logarithm transformation of the number of weeks on treatment was included as an offset variable in the model; Test type: Superiority; p = 0.1335, Modified Poisson — [p-value comment as in outcome 1, analysis 1]; Hochberg-based gatekeeping procedure

5. Secondary Outcome: Occurrence of Granulocyte Colony-Stimulating Factor (G-CSF) Administration (Proportion of Patients)
Description: For this endpoint, the occurrence during the Induction Period was defined as a binary variable (Yes or No); Yes, if total number of events ≥1 was observed, No for other scenarios. If a patient did not have an event, a value of 0 was assigned to that patient. Any G-CSF administration in a cycle during the Induction Period was defined as a separate event. A patient with at least 1 cycle with G-CSF administration during an induction cycle or the Induction Period was considered to have occurrence of G-CSF administration.
Time Frame: as for outcome 3
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Trilaciclib+Etoposide/Carboplatin/Atezolizumab | Placebo+Etoposide/Carboplatin/Atezolizumab
Number analyzed (Participants) | 54 | 53
Participants | 16 | 25
Statistical Analysis 1: Comparison: Trilaciclib+Etoposide/Carboplatin/Atezolizumab vs Placebo+Etoposide/Carboplatin/Atezolizumab; Treatment group difference was analyzed using a modified Poisson regression model to account for the variable duration of the Induction Period for each patient. The model included baseline absolute neutrophil count as a covariate, the stratification factors of ECOG performance status (0 to 1 versus 2) and brain metastases (Yes versus No), and treatment as a fixed effect. The logarithm transformation of number of Induction cycles was included as an offset variable in the modeling; Test type: Superiority; p = 0.0686, Modified Poisson — [p-value comment as in outcome 1, analysis 1]; Hochberg-based gatekeeping procedure

6. Secondary Outcome: Overall Survival (OS)
Description: Overall survival was calculated as the time (months) from date of randomization to the date of death due to any cause. Patients who did not die during the study were censored at the date last known to be alive. Patients lacking data beyond the date of randomization had their survival time censored at date of randomization. Overall survival was not censored if a patient received other anti-tumor treatments after the study drugs. Overall survival was calculated using the Kaplan-Meier method.
Time Frame: From date of randomization to date of death due to any cause, assessed up to a maximum of 38.1 months.
Population: Intent-to-treat (ITT Analysis Set)
Measure: Number (95% Confidence Interval); unit: Months
Groups:
- Trilaciclib+Etoposide/Carboplatin/Atezolizumab: Induction: Patients received trilaciclib 240 mg/m² administered IV once daily prior to E/P/A on Days 1, 2 and 3 of each 21-day E/P/A therapy cycle (up to 4 cycles in total). Etoposide 100 mg/m² was administered IV daily on Days 1, 2, and 3 of each 21-day cycle. Carboplatin was administered on Day 1 of each 21-day cycle using the Calvert formula with a target AUC = 5 mg/mL/min to calculate the dose. Atezolizumab 1200 mg was administered as an IV infusion on Day 1 of each 21-day cycle.
  Maintenance: Following the induction phase, patients received maintenance atezolizumab at a dose of 1200 mg on Day 1 of every 21-day cycle until disease progression, unacceptable toxicity or discontinuation by the patient or investigator.
Arm/Group | Trilaciclib+Etoposide/Carboplatin/Atezolizumab | Placebo+Etoposide/Carboplatin/Atezolizumab
Number analyzed (Participants) | 54 | 53
Months
  25% | 7.2 [4.9 to 10.2] | 6.7 [3.6 to 8.1]
  Median | 12.0 [9.6 to 16.2] | 12.8 [7.9 to 15.5]
  75% | 20.6 [14.5 to 23.2] | 22.4 [15.5 to 30.0]
Statistical Analysis 1: Comparison: Trilaciclib+Etoposide/Carboplatin/Atezolizumab vs Placebo+Etoposide/Carboplatin/Atezolizumab; Test type: Superiority — For time-to-event variable, the Kaplan-Meier method was used to estimate its within group median value, 25% and 75% percentile values; p = 0.9942, Log Rank — The 2-sided p-value was obtained from the stratified log-rank test to account for the stratification factors; stratified log-rank test; Hazard Ratio (HR) = 0.99, 95% CI 2-sided [0.64 to 1.52], Standard Error of Mean 0.218 — The HR and its 95% CI were calculated using the Cox proportional hazard regression model with treatment and stratification factors of ECOG performance status (0 to 1 versus 2) and presence of brain metastases (Yes versus No)

7. Secondary Outcome: Major Adverse Hematologic Events (MAHE) (Composite Endpoint)
Description: The composite endpoint "major adverse hematologic events" (MAHE) included the following aspects of myelosuppression:
  All-cause hospitalizations - Each recorded preferred term (PT) with a unique start date was counted as an event.
  All-cause dose reductions - Dose reductions were permitted for E/P but not for trilaciclib or atezolizumab. No more than 2 dose reductions were allowed. Each dose reduction was counted as a separate event.
  Febrile neutropenia-Each febrile neutropenia event with a unique start date during the Induction Period was defined as a separate event.
  Prolonged severe neutropenia (SN)-Each cycle with a severe neutropenia duration greater than 5 days was counted as an event, with the date of the first Grade 4 laboratory value defined as the start date for the time-to-first event analysis.
  Red blood cell (RBC) transfusion on/after Week 5-Each RBC transfusion with a unique start date on/after Week 5 on study during the Induction Period was defined as a separate event.
Time Frame: as for outcome 3
Population: as for outcome 1
Measure: Number; unit: event rate per week
Arm/Group | Trilaciclib+Etoposide/Carboplatin/Atezolizumab | Placebo+Etoposide/Carboplatin/Atezolizumab
Number analyzed (Participants) | 54 | 53
event rate per week
  Major adverse hematologic events (MAHE) | 0.132 | 0.058
  All-cause hospitalizations | 0.032 | 0.030
  All-cause dose reductions | 0.021 | 0.085
  Febrile neutropenia TEAEs | 0.002 | 0.004
  RBC transfusions on/after Week 5 | 0.017 | 0.026
  Prolonged SN (>5 days) | 0.005 | 0.170

8. Secondary Outcome: Best Overall Response
Description: For all patients, the Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) tumor response data were used to determine each patient's visit response (TPR = time point response). Per RECIST v1.1 for target lesions and assessed by CT/MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameters of target lesions; Progressive Disease (PD), >=20% increase in the sum of the longest diameter of target lesions, Stable Disease, neither sufficient shrinkage or increase to quality for PR or PD. Objective Response Rate (ORR) = CR + PR. The TPR at each visit was determined in 2 ways: (1) derived programmatically at the time of analysis using the information from target lesions, non-target lesions, and new lesions based on data collected through eCRF; and (2) judged by the investigator as collected in the eCRF. Results shown here are from the programmatically derived assessments.
Time Frame: From date of randomization, up to four 21-day cycles of Induction therapy, followed by 21 day cycles of Maintenance therapy until disease progression, unacceptable toxicity or discontinuation by the patient or investigator, assessed up to 724 days.
Population: Response Evaluable Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Trilaciclib+Etoposide/Carboplatin/Atezolizumab | Placebo+Etoposide/Carboplatin/Atezolizumab
Number analyzed (Participants) | 50 | 52
Participants
  Complete Response (CR) | 0 | 1
  Partial Response (PR) | 28 | 32
  Stable Disease (SD) | 20 | 14
  Progressive Disease (PD) | 2 | 2
  Not Evaluable (NE) | 0 | 2
  Missing | 0 | 1
  Objective response rate (CR+PR) | 28 | 33

9. Secondary Outcome: Duration of Objective Response (Complete Response or Partial Response)
Description: Duration of Response (DOR) is the time between first response by RECIST Version 1.1 of CR or PR and the first date that progressive disease is documented by RECIST Version 1.1, or death. Patients who do not experience PD or death will be censored at the last tumor assessment date. Only those patients with confirmed responses will be included in this analysis.
Time Frame: as for outcome 8
Population: Response Evaluable Analysis Set
Measure: Number (95% Confidence Interval); unit: months
Arm/Group | Trilaciclib+Etoposide/Carboplatin/Atezolizumab | Placebo+Etoposide/Carboplatin/Atezolizumab
Number analyzed (Participants) | 28 | 33
months
  25% | 4.4 [2.9 to 4.7] | 3.0 [2.7 to 4.1]
  Median | 5.6 [4.4 to 7.0] | 4.3 [3.4 to 4.7]
  75% | 8.3 [5.8 to 13.2] | 5.0 [4.6 to 10.5]

10. Secondary Outcome: Progression-Free Survival
Description: Progression-free survival (PFS) was defined as the time (number of months) from date of randomization until date of documented radiologic disease progression per RECIST v1.1 or death due to any cause, whichever came first.
Time Frame: as for outcome 8
Population: Intent-to-treat
Measure: Number (95% Confidence Interval); unit: months
Arm/Group | Trilaciclib+Etoposide/Carboplatin/Atezolizumab | Placebo+Etoposide/Carboplatin/Atezolizumab
Number analyzed (Participants) | 54 | 53
months
  25% | 3.7 [2.7 to 4.2] | 4.0 [3.1 to 4.3]
  Median | 5.9 [4.2 to 7.1] | 5.4 [4.3 to 5.7]
  75% | 8.5 [7.1 to 10.4] | 6.4 [5.7 to 8.9]

11. Secondary Outcome: Number of Participants With at Least 1 Occurrence of Febrile Neutropenia
Description: The criterion for identifying febrile neutropenia was if the preferred term for an adverse event was "FEBRILE NEUTROPENIA." Any occurrence of a febrile neutropenia event during the induction treatment period is defined as a binary variable (Yes or No); Yes if total number of febrile neutropenia events ≥ 1 is observed, No for other scenarios. Each febrile neutropenia event with a unique start date during the induction treatment period was defined as a separate event.
Time Frame: as for outcome 3
Population: Intent-to-treat (ITT Analysis Set)
Measure: Count of Participants; unit: Participants
Arm/Group | Trilaciclib+Etoposide/Carboplatin/Atezolizumab | Placebo+Etoposide/Carboplatin/Atezolizumab
Number analyzed (Participants) | 54 | 53
Participants | 1 | 3

12. Secondary Outcome: Number of Participants With at Least 1 Occurrence of Grade 3 or 4 Hematologic Laboratory Abnormalities
Description: The occurrence of Grade 3 and 4 hematologic toxicities was a binary endpoint. If a patient had at least 1 cycle with at least 1 Grade 3 or 4 hematologic toxicities during the Induction Period, the patient was assigned as "Yes" to the occurrence of Grade 3 and 4 hematologic toxicities; otherwise, it was "No". If a patient did not have an event, the value of 0 was assigned to that patient.
Time Frame: as for outcome 3
Population: Intent-to-treat
Measure: Count of Participants; unit: Participants
Arm/Group | Trilaciclib+Etoposide/Carboplatin/Atezolizumab | Placebo+Etoposide/Carboplatin/Atezolizumab
Number analyzed (Participants) | 54 | 53
Participants | 23 | 43

13. Secondary Outcome: Number of Participants With at Least 1 Occurrence of Erythropoiesis Stimulating Agent (ESA) Administration
Description: Any ESA administration in a cycle during the Induction Period was defined as a separate event. A patient with at least 1 cycle with ESA administration during an induction cycle or the Induction Period was considered to have occurrence of ESA administration. The criterion to select proper records was as follows: If the chemical subgroup from WHO-DD Version September 2017 (ie TEXT4 for CODE4) takes the value "OTHER ANTIANEMIC PREPARATIONS," the medication was classified as ESAs.
Time Frame: as for outcome 3
Population: Intent-to-treat
Measure: Count of Participants; unit: Participants
Arm/Group | Trilaciclib+Etoposide/Carboplatin/Atezolizumab | Placebo+Etoposide/Carboplatin/Atezolizumab
Number analyzed (Participants) | 54 | 53
Participants | 3 | 6

14. Secondary Outcome: Number of Participants With at Least 1 Occurrence of Platelet Transfusion
Description: Any occurrence of a platelet transfusion during the induction treatment period was defined as a binary variable (Yes or No); Yes if total number of febrile neutropenia events ≥ 1 is observed, No for other scenarios. If the patient did not have an event, the value of 0 was assigned to that patient. Each platelet transfusion event with a unique start date during the induction treatment period was defined as a separate event.
Time Frame: as for outcome 3
Population: Intent-to-treat
Measure: Count of Participants; unit: Participants
Arm/Group | Trilaciclib+Etoposide/Carboplatin/Atezolizumab | Placebo+Etoposide/Carboplatin/Atezolizumab
Number analyzed (Participants) | 54 | 53
Participants | 1 | 2

15. Secondary Outcome: Number of Participants With at Least 1 Occurrence of Infection Serious Adverse Events (SAEs)
Description: Any occurrence of an infection SAE during the induction treatment period was defined as a binary variable (Yes or No); Yes if total number of febrile neutropenia events ≥ 1 is observed, No for other scenarios. If the patient did not have an event, the value of 0 was assigned to that patient. The criterion for identifying the proper infection SAE records was as follows: if the system organ class (SOC) from Medical Dictionary for Regulatory Activities (MedDRA) Version 20.1 takes value "INFECTIONS AND INFESTATIONS," and the AE was a serious event.
Time Frame: as for outcome 3
Population: Intent-to-treat
Measure: Count of Participants; unit: Participants
Arm/Group | Trilaciclib+Etoposide/Carboplatin/Atezolizumab | Placebo+Etoposide/Carboplatin/Atezolizumab
Number analyzed (Participants) | 54 | 53
Participants | 3 | 7

16. Secondary Outcome: Number of Participants With at Least 1 Occurrence of Pulmonary Infection Serious Adverse Events (SAEs)
Description: Any occurrence of a pulmonary SAE during the induction treatment period was defined as a binary variable (Yes or No); Yes if total number of febrile neutropenia events ≥ 1 is observed, No for other scenarios. If the patient did not have an event, the value of 0 was assigned to that patient. Each pulmonary infection SAE with a unique start date during the induction treatment period was defined as separate event. The criterion for identifying the proper pulmonary infection SAE records was as follows:
  The SOC from MedDRA Version 20.1 took the value "INFECTIONS AND INFESTATIONS," the adverse event was a serious event, and the PT took values from the following list of PTs under the category of pulmonary infection adverse events: bronchiolitis, bronchitis, infectious pleural effusion, influenza, pneumonia, pneumonia bacterial, respiratory tract infection, upper respiratory tract infection, and viral upper respiratory tract infection.
Time Frame: as for outcome 3
Population: Intent-to-treat
Measure: Count of Participants; unit: Participants
Groups:
- Placebo+Etoposide/Carboplatin/Atezolizumab: Induction: Patients will receive placebo administered IV once daily prior to E/P/A on Days 1, 2 and 3 of each 21-day E/P/A therapy cycle (up to 4 cycles in total). Etoposide 100 mg/m² will be administered IV daily on Days 1, 2, and 3 of each 21-day cycle. Carboplatin will be administered on Day 1 of each 21-day cycle using the Calvert formula with a target AUC = 5 mg/mL/min to calculate the dose. Atezolizumab 1200 mg will be administered as an IV infusion on Day 1 of each 21-day cycle.
  Maintenance: Following the induction phase, patients will receive maintenance atezolizumab at a dose of 1200 mg on Day 1 of every 21-day cycle until disease progression, unacceptable toxicity, or discontinuation by the patient or investigator.
Arm/Group | Trilaciclib+Etoposide/Carboplatin/Atezolizumab | Placebo+Etoposide/Carboplatin/Atezolizumab
Number analyzed (Participants) | 54 | 53
Participants | 2 | 5

17. Secondary Outcome: Number of Participants With at Least 1 Occurrence of IV Antibiotic Uses
Description: Occurrence of an IV antibiotics administration during the induction treatment period is defined as a binary variable (Yes or No); Yes if total number of IV antibiotics administration ≥ 1 is observed, No for other scenarios. Each IV antibiotic with a unique start date during the induction treatment period will be defined as a separate event. The criteria for identifying an IV antibiotic administration event was (1) if the therapeutic subgroup from WHO-DD Version September 2017 (ie, TEXT2 for CODE2) takes the value "ANTIBACTERIALS FOR SYSTEMIC USE," and (2) the route of medication was "intravenous" or the route was "other" with the detailed specification as "IVPB."
Time Frame: as for outcome 3
Population: Intent-to-treat
Measure: Count of Participants; unit: Participants
Groups:
- Placebo+Etoposide/Carboplatin/Atezolizumab: Induction: Patients received placebo administered IV once daily prior to E/P/A on Days 1, 2 and 3 of each 21-day E/P/A therapy cycle (up to 4 cycles in total). Etoposide 100 mg/m2 was administered IV daily on Days 1, 2, and 3 of each 21-day cycle. Carboplatin was administered on Day 1 of each 21-day cycle using the Calvert formula with a target AUC = 5 mg/mL/min to calculate the dose. Atezolizumab 1200 mg was administered as an IV infusion on Day 1 of each 21-day cycle.
  Maintenance: Following the induction phase, patients received maintenance atezolizumab at a dose of 1200 mg on Day 1 of every 21-day cycle until disease progression, unacceptable toxicity, or discontinuation by the patient or investigator.
Arm/Group | Trilaciclib+Etoposide/Carboplatin/Atezolizumab | Placebo+Etoposide/Carboplatin/Atezolizumab
Number analyzed (Participants) | 54 | 53
Participants | 10 | 12

18. Secondary Outcome: Duration of Study Drug Exposure (Induction Period and Maintenance Period)
Description: Induction period duration of exposure (days) = Day 1 of last induction cycle - Cycle 1 Day 1 of induction phase + 21. Maintenance period duration of exposure (days) = Day 1 of the last maintenance cycle -Cycle 1 Day 1 of maintenance phase + 21.
Time Frame: From date of first dose, up to four 21-day cycles of Induction therapy, followed by 21 day cycles of Maintenance therapy until disease progression, unacceptable toxicity or discontinuation by the patient or investigator, assessed up to 1162 days.
Population: Safety analysis
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Trilaciclib+Etoposide/Carboplatin/Atezolizumab | Placebo+Etoposide/Carboplatin/Atezolizumab
Number analyzed (Participants) | 52 | 53
Days
  Induction Period | 83 (15.6) | 88 (20.5)
  Maintenance Period: number analyzed (Participants) | 41 | 47
  Maintenance Period | 223 (253.3) | 232 (271.0)

19. Secondary Outcome: Number of Cycles Completed (Induction Period and Maintenance Period)
Description: Patients were considered to have started a cycle if they have received at least one dose of any study drug (carboplatin, etoposide, atezolizumab or trilaciclib).
Time Frame: From date of first dose, up to four 21-day cycles of Induction therapy, followed by 21 day cycles of Maintenance therapy until disease progression, unacceptable toxicity or discontinuation by the patient or investigator, assessed up to 49 cycles.
Population: Safety analysis
Measure: Mean (Standard Deviation); unit: Cycles
Arm/Group | Trilaciclib+Etoposide/Carboplatin/Atezolizumab | Placebo+Etoposide/Carboplatin/Atezolizumab
Number analyzed (Participants) | 52 | 53
Cycles
  Induction Period | 4 (0.6) | 4 (0.8)
  Maintenance Period: number analyzed (Participants) | 41 | 47
  Maintenance Period | 10 (11.9) | 10 (11.3)

20. Secondary Outcome: Relative Dose Intensity of Trilaciclib/Placebo, Carboplatin, Etoposide, Atezolizumab (Induction Period) and Atezolizumab (Maintenance Period)
Description: Relative dose intensity is defined as 100% times the actual dose intensity divided by the planned dose intensity. The planned dose intensity is defined as the cumulative planned dose through the study divided by (number of cycles * 3 weeks)
Time Frame: From date of first dose, up to four 21-day cycles of Induction therapy, followed by 21 day cycles of Maintenance therapy until disease progression, unacceptable toxicity or discontinuation by the patient or investigator, assessed up to 724 days.
Population: Safety Analysis
Measure: Mean (Standard Deviation); unit: percentage of dose
Arm/Group | Trilaciclib+Etoposide/Carboplatin/Atezolizumab | Placebo+Etoposide/Carboplatin/Atezolizumab
Number analyzed (Participants) | 52 | 53
percentage of dose
  Trilaciclib/Placebo | 94.6 (7.65) | 91.1 (10.68)
  Carboplatin | 95.3 (7.65) | 89.1 (12.25)
  Etoposide | 93.4 (9.59) | 87.7 (13.92)
  Atezolizumab (Induction) | 94.1 (9.54) | 91.0 (11.26)
  Atezolizumab (Maintenance) | 93.5 (11.45) | 94.2 (10.19)

21. Secondary Outcome: Number of Participants With Any Cycle Delays and the Number of Cycles Delayed (Induction Period)
Description: After Cycle 1, patients need to meet pre-specified laboratory parameter criteria before initiating Cycle 2 and each subsequent cycle of chemotherapy. A "Cycle Day Status" page asks if the cycle was delayed. If the start of the current cycle was delayed (the site answers "Yes"), this will be counted as a delay. Cycle delays could occur for management of toxicity (hematologic or non-hematologic) or for administrative/logistic reasons. The reason for each cycle delay was captured in the eCRF if it was related to AEs. Reasons other than AEs were not captured.
Time Frame: Induction Period. From date of first dose, 21 day treatment cycles to a maximum of 4 cycles or until (if earlier) disease progression, unacceptable toxicity, or discontinuation by the patient or investigator, assessed up to a maximum of 409 days.
Population: Safety analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Trilaciclib+Etoposide/Carboplatin/Atezolizumab | Placebo+Etoposide/Carboplatin/Atezolizumab
Number analyzed (Participants) | 52 | 53
Participants
  Number of patients with any cycle delays | 18 | 31
  0 cycles | 34 | 22
  1 cycle | 14 | 18
  2 cycles | 2 | 10
  3 or more cycles | 2 | 3

22. Secondary Outcome: Number of Participants With Any Cycle Delays and the Number of Cycles Delayed (Maintenance Period)
Description: as for outcome 21
Time Frame: Maintenance Period. From date of first maintenance dose, 21 day cycles of Maintenance therapy until disease progression, unacceptable toxicity or discontinuation by the patient or investigator, assessed up to 1160 days.
Population: Safety analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Trilaciclib+Etoposide/Carboplatin/Atezolizumab | Placebo+Etoposide/Carboplatin/Atezolizumab
Number analyzed (Participants) | 52 | 53
Participants
  Number of patients with any cycle delays | 21 | 26
  0 cycles | 20 | 21
  1 cycle | 10 | 12
  2 cycles | 6 | 6
  3 or more cycles | 5 | 8

23. Secondary Outcome: Number of Participants With Any Missed Doses [for Each Study Drug: Trilaciclib/Placebo, Carboplatin and Etoposide] (Induction Period)
Description: Missed doses are identified on the dosing page of each study drug based on the question "Was the dose given?". The missed dose information will be obtained for each study drug. For a study drug, if the last record of response to question "Was the dose given?" is No, it will not be considered as a missed dose but instead considered to be end of treatment if both criteria below are met: (1) No other study drugs are given on the same day, and (2) No study drugs are given subsequently.
Time Frame: as for outcome 21
Population: Safety analysis
Measure: Count of Participants; unit: Participants
Groups:
- Placebo+Etoposide/Carboplatin/Atezolizumab: Induction: Patients received placebo administered IV once daily prior to E/P/A on Days 1, 2 and 3 of each 21-day E/P/A therapy cycle (up to 4 cycles in total). Etoposide 100 mg/m² was administered IV daily on Days 1, 2, and 3 of each 21-day cycle. Carboplatin was administered on Day 1 of each 21-day cycle using the Calvert formula with a target AUC = 5 mg/mL/min to calculate the dose. Atezolizumab 1200 mg was administered as an IV infusion on Day 1 of each 21-day cycle.
  Maintenance: Following the induction phase, patients receives maintenance atezolizumab at a dose of 1200 mg on Day 1 of every 21-day cycle until disease progression, unacceptable toxicity, or discontinuation by the patient or investigator.
Arm/Group | Trilaciclib+Etoposide/Carboplatin/Atezolizumab | Placebo+Etoposide/Carboplatin/Atezolizumab
Number analyzed (Participants) | 52 | 53
Participants
  Trilaciclib/Placebo | 3 | 0
  Carboplatin | 1 | 0
  Etoposide | 3 | 0

24. Secondary Outcome: Number of Participants With Any Missed Doses of Atezolizumab (Overall Treatment Period)
Description: as for outcome 23
Time Frame: as for outcome 18
Population: Safety analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Trilaciclib+Etoposide/Carboplatin/Atezolizumab | Placebo+Etoposide/Carboplatin/Atezolizumab
Number analyzed (Participants) | 52 | 53
Participants | 3 | 3

25. Secondary Outcome: Number of Participants With Any Dose Interruptions [for Each Study Drug: Trilaciclib/Placebo, Carboplatin and Etoposide] (Induction Period)
Description: Dose interruptions were defined as interruption of infusion, regardless of whether the study drug was continued after the interruption.
Time Frame: as for outcome 21
Population: Safety analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Trilaciclib+Etoposide/Carboplatin/Atezolizumab | Placebo+Etoposide/Carboplatin/Atezolizumab
Number analyzed (Participants) | 52 | 53
Participants
  Trilaciclib/placebo | 3 | 0
  Carboplatin | 0 | 1
  Etoposide | 2 | 3

26. Secondary Outcome: Number of Participants With Any Interrupted Doses of Atezolizumab (Overall Treatment Period)
Description: as for outcome 25
Time Frame: as for outcome 18
Population: Safety analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Trilaciclib+Etoposide/Carboplatin/Atezolizumab | Placebo+Etoposide/Carboplatin/Atezolizumab
Number analyzed (Participants) | 52 | 53
Participants | 1 | 0

27. Secondary Outcome: Number of Participants With Any Dose Reductions of Carboplatin and Etoposide (Induction Period)
Description: No dose reductions were allowed for trilaciclib or atezolizumab during the study.
Time Frame: as for outcome 21
Population: Safety analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Trilaciclib+Etoposide/Carboplatin/Atezolizumab | Placebo+Etoposide/Carboplatin/Atezolizumab
Number analyzed (Participants) | 52 | 53
Participants
  Etoposide | 3 | 14
  Carboplatin | 1 | 13

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events collected beginning with informed consent through 30 days after last dose of study drug. Treatment emergent serious adverse events collected through 90 days after last dose of study drug, assessed up to a maximum of 1192 days (maximum duration of exposure plus 30 days).
Description: Adverse events were assessed using the safety analysis set, which included all randomized patients who received at least 1 dose of any study drug (etoposide, carboplatin, atezolizumab, or trilaciclib). Analyses using the safety analysis set were conducted based on the actual treatment received.
Arm/Group | Trilaciclib+Etoposide/Carboplatin/Atezolizumab | Placebo+Etoposide/Carboplatin/Atezolizumab
All-Cause Mortality (participants affected / at risk) | 42/54 | 44/53
Serious Adverse Events (participants affected / at risk) | 17/52 | 25/53
Other Adverse Events (participants affected / at risk) | 49/52 | 52/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Trilaciclib+Etoposide/Carboplatin/Atezolizumab (N=52) | Placebo+Etoposide/Carboplatin/Atezolizumab (N=53)
Pneumonia (Infections and infestations) | 3 (5) | 8 (8)
Sepsis (Infections and infestations) | 0 (0) | 2 (2)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 1 (1)
Bronchiolitis (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Empyema (Infections and infestations) | 0 (0) | 1 (2)
Meningoencephalitis herpetic (Infections and infestations) | 0 (0) | 1 (2)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 4 (4)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 3 (3)
Anaemia (Blood and lymphatic system disorders) | 1 (2) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 1 (1)
Balance disorder (Nervous system disorders) | 0 (0) | 1 (1)
Cognitive disorder (Nervous system disorders) | 0 (0) | 1 (1)
Generalised tonic-clonic seizure (Nervous system disorders) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Paraneoplastic neurological syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1) | 1 (1)
Asthenia (General disorders) | 0 (0) | 1 (2)
Oedema peripheral (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (5) | 2 (2)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 1 (1) | 0 (0)
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1)
Angioedema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Trilaciclib+Etoposide/Carboplatin/Atezolizumab (N=52) | Placebo+Etoposide/Carboplatin/Atezolizumab (N=53)
Anaemia (Blood and lymphatic system disorders) | 19 (60) | 32 (122)
Neutropenia (Blood and lymphatic system disorders) | 19 (35) | 28 (85)
Thrombocytopenia (Blood and lymphatic system disorders) | 7 (14) | 21 (44)
Leukopenia (Blood and lymphatic system disorders) | 4 (5) | 14 (38)
Fatigue (General disorders) | 16 (24) | 20 (32)
Asthenia (General disorders) | 8 (17) | 9 (21)
Non-cardiac chest pain (General disorders) | 5 (5) | 7 (7)
Pyrexia (General disorders) | 8 (8) | 4 (5)
Oedema peripheral (General disorders) | 4 (4) | 4 (4)
Chills (General disorders) | 2 (2) | 4 (5)
Gait disturbance (General disorders) | 1 (1) | 3 (3)
Nausea (Gastrointestinal disorders) | 20 (36) | 18 (30)
Constipation (Gastrointestinal disorders) | 5 (6) | 12 (15)
Diarrhoea (Gastrointestinal disorders) | 9 (13) | 6 (10)
Vomiting (Gastrointestinal disorders) | 6 (10) | 5 (6)
Stomatitis (Gastrointestinal disorders) | 3 (3) | 3 (5)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 4 (5)
Dyspepsia (Gastrointestinal disorders) | 4 (4) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 7 (8) | 18 (21)
Pruritus (Skin and subcutaneous tissue disorders) | 8 (9) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 5 (10) | 4 (5)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (11)
Platelet count decreased (Investigations) | 5 (10) | 13 (63)
Neutrophil count decreased (Investigations) | 3 (11) | 11 (50)
White blood cell count decreased (Investigations) | 7 (20) | 6 (25)
Aspartate aminotransferase increased (Investigations) | 6 (11) | 2 (4)
Alanine aminotransferase increased (Investigations) | 5 (10) | 2 (4)
Blood alkaline phosphatase increased (Investigations) | 4 (5) | 3 (6)
Blood creatinine increased (Investigations) | 3 (4) | 4 (5)
Blood lactate dehydrogenase increased (Investigations) | 3 (5) | 4 (8)
Weight decreased (Investigations) | 4 (5) | 3 (3)
Lipase increased (Investigations) | 1 (2) | 5 (10)
Weight increased (Investigations) | 3 (3) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 (13) | 13 (20)
Cough (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 8 (12)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 5 (7)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (4)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Urinary tract infection (Infections and infestations) | 5 (7) | 3 (4)
Pneumonia (Infections and infestations) | 4 (4) | 3 (4)
Upper respiratory tract infection (Infections and infestations) | 3 (4) | 3 (5)
Bronchitis (Infections and infestations) | 3 (4) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 5 (6) | 9 (11)
Decreased appetite (Metabolism and nutrition disorders) | 4 (5) | 9 (10)
Hyperglycaemia (Metabolism and nutrition disorders) | 5 (11) | 3 (3)
Hyponatraemia (Metabolism and nutrition disorders) | 4 (13) | 4 (4)
Hypokalaemia (Metabolism and nutrition disorders) | 4 (6) | 2 (2)
Hyperkalaemia (Metabolism and nutrition disorders) | 3 (7) | 1 (1)
Dizziness (Nervous system disorders) | 9 (11) | 9 (13)
Headache (Nervous system disorders) | 9 (13) | 6 (9)
Tremor (Nervous system disorders) | 1 (1) | 3 (3)
Dysgeusia (Nervous system disorders) | 0 (0) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (10) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (5) | 2 (2)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (3)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (4)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3)
Hypertension (Vascular disorders) | 3 (6) | 3 (4)
Flushing (Vascular disorders) | 3 (4) | 2 (2)
Hypotension (Vascular disorders) | 1 (1) | 3 (4)
Phlebitis (Vascular disorders) | 3 (4) | 0 (0)
Hypothyroidism (Endocrine disorders) | 3 (3) | 7 (7)
Hyperthyroidism (Endocrine disorders) | 2 (3) | 6 (6)
Anxiety (Psychiatric disorders) | 3 (8) | 5 (5)
Confusional state (Psychiatric disorders) | 2 (2) | 4 (5)
Insomnia (Psychiatric disorders) | 0 (0) | 4 (4)
Urinary incontinence (Renal and urinary disorders) | 1 (4) | 3 (5)
Infusion related reaction (Injury, poisoning and procedural complications) | 5 (11) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 2 (3) | 4 (6)

LIMITATIONS AND CAVEATS:
Limitation of the trial is small numbers of subjects, since it is a Phase 2 clinical trial.

Small sample size may have reduced the ability to observe statistically significant treatment effects on secondary myelopreservation measures (i.e. occurrence of FN AEs, infections and antibiotics usage).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2018-09-14): https://cdn.clinicaltrials.gov/large-docs/11/NCT03041311/Prot_000.pdf
  • Statistical Analysis Plan: Region 2 (2018-11-01): https://cdn.clinicaltrials.gov/large-docs/11/NCT03041311/SAP_001.pdf